CLINICAL TRIAL: NCT05836389
Title: Long-term Results of Bilateral Thoracoscopic Ablation for Stand-alone Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of the Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: LTFUP-AFPVI
Record Dates: First submitted 2023-01-27; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pulmonary veins isoltation in bilateral thoracoscopy — Ablation of the atrial fibrillation performin isolation of the pulmonary vein. The procedure is video-assisted, access is minimally invasive: access to the heart is provided to instruments and camera via small bilateral chest incisions

SUMMARY:
Atrial fibrillation (AFib) represents the most frequent cardiac arrhythmia whose prevalence appears to be increasing in the general population. Furthermore, this arrhythmia determines an increased risk of neurological complications (stroke) and, consequently, of mortality and morbidity.

Currently, the first choice for the treatment of AFib is represented by the use of antiarrhythmic drugs. In patients who do not respond to pharmacological treatment, the ESC 2016 European guidelines recommend the execution of transcatheter ablation (Class I, level of evidence A). However, minimally invasive pulmonary vein isolation surgery (PVI) is recommended for subjects who are not even responsive to transcatheter ablation (Class IIa, Level of Evidence B).

Previous studies have demonstrated good short-term results of thoracoscopic AFib ablation using PVI, with a 1-year freedom from atrial fibrillation recurrence without antiarrhythmic drugs of approximately 64-73%. However, only a few authors have described the medium-long term follow-up outcomes.

The aim of this study is to report the long-term follow-up data of ablation of isolated, predominantly paroxysmal atrial fibrillation performed by isolation of the pulmonary veins by radiofrequency in bilateral thoracoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years old;
* Isolated atrial fibrillation (predominantly paroxysmal);
* Patients undergoing ablation of atrial fibrillation (both paroxysmal and persistent) by isolation of the pulmonary veins by radiofrequency in thoracoscopy.

Exclusion Criteria:

* Age under 20 or over 80;
* Previous trauma/deformity of the rib cage limiting the thoracoscopic approach;
* Previous pleurisy or thoracic operations (e.g. lobectomies) conditioning the possible appearance of pleural adhesions limiting the thoracoscopic approach.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent isolated ablation of paroxysmal or persistent AFib with pulmonary veins isolation in bilateral thoracoscopy
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, a minimum of 6 years
Freedom from AFib | through study completion, a minimum of 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No